CLINICAL TRIAL: NCT02725268
Title: A Phase 2, Randomized Study of MLN0128 (a Dual TORC1/2 Inhibitor), MLN0128+MLN1117 (a PI3Kα Inhibitor), Weekly Paclitaxel, or the Combination of Weekly Paclitaxel and MLN0128 in Women With Advanced, Recurrent, or Persistent Endometrial Cancer
Brief Title: A Study of Sapanisertib, Combination of Sapanisertib With MLN1117, Paclitaxel and Combination of Sapanisertib With Paclitaxel in Women With Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: European Network of Translational Research in Ovarian Cancer - EUTROC (Unknown); European Network of Individualized Treatment in Endometrial Cancer - ENITEC (Other Government)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C31004; U1111-1168-1824 (Other: WHO); 2014-005394-37 (EudraCT Number); 02725268 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Endometrial Neoplasms
Keywords: Drug Therapy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel; sapanisertib; serabelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Paclitaxel 80 mg/m^2 (Experimental): Paclitaxel 80 milligrams per square meter (mg/m^2), IV, weekly on Days 1, 8, and 15 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was up to approximately 13 weeks).
  Interventions: Drug: Paclitaxel
- Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg (Experimental): Paclitaxel 80 mg/m^2, IV, weekly on Days 1, 8, and 15 of a 28-day cycle along with sapanisertib 4 milligrams (mg), capsule, orally on Days 2-4, 9-11, 16-18, and 23-25 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was up to approximately 20 weeks).
  Interventions: Drug: Paclitaxel; Drug: Sapanisertib
- Sapanisertib 30 mg (Experimental): Sapanisertib 30 mg, capsule, orally, once weekly on Days 1, 8, 15, and 22 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was up to approximately 6 weeks).
  Interventions: Drug: Sapanisertib
- Sapanisertib 4 mg + MLN1117 200 mg (Experimental): Sapanisertib 4 mg, capsule, orally and MLN1117 200 mg, capsule, orally on Days 1-3, 8-10, 15-17, and 22-24 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was up to approximately 8 weeks).
  Interventions: Drug: Sapanisertib; Drug: MLN1117

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel intravenous solution.
  Arms: Paclitaxel 80 mg/m^2; Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg
Drug: Sapanisertib — Sapanisertib capsules.
  Other Names: MLN0128; INK128; TAK-228
  Arms: Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg; Sapanisertib 30 mg; Sapanisertib 4 mg + MLN1117 200 mg
Drug: MLN1117 — MLN1117 capsules.
  Other Names: TAK-117; INK1117
  Arms: Sapanisertib 4 mg + MLN1117 200 mg

SUMMARY:
The primary purpose of this study is to determine if sapanisertib in combination with weekly paclitaxel improves progression-free survival (PFS) compared to weekly paclitaxel alone.

DETAILED DESCRIPTION:
The drugs being evaluated in this study are sapanisertib and MLN1117. Sapanisertib is being evaluated as a single agent and in combination with paclitaxel or MLN1117 to treat women with advanced, recurrent, or persistent endometrial cancer. This study will evaluate the efficacy and safety of each drug or drug combination.

The study will enroll approximately 241 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of 4 treatment groups:

* Paclitaxel 80 mg/m^2
* Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg
* Sapanisertib 30 mg
* Sapanisertib 4 mg + MLN1117 200 mg

Participants will receive either paclitaxel intravenous (IV) weekly, Paclitaxel IV along with sapanisertib orally, sapanisertib orally, or sapanisertib and MLN1117 orally.

This is a multicenter, multinational trial. Participants will make multiple visits to the clinic, with an end of treatment visit (EOT) which will occur 30 to 40 days after receiving their last dose of study drug or before the start of any subsequent anticancer therapy. After EOT, participants will be followed for PFS and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of endometrial carcinoma (including endometrioid, serous, mixed adenocarcinoma, clear-cell carcinoma, or carcinosarcoma).
2. Evidence that the endometrial cancer is advanced, recurrent, or persistent and has relapsed or is refractory to curative therapy or established treatments.
3. At least 1 prior platinum-based chemotherapeutic regimen, but not more than 2 prior chemotherapeutic regimens, for management of endometrial carcinoma. Prior treatment may include chemotherapy, chemotherapy/radiation therapy, and/or consolidation/maintenance therapy. Chemotherapy administered in conjunction with primary radiation as a radio-sensitized therapy will be considered a systemic chemotherapy regimen.
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded). Each lesion must be greater than or equal to (>=) 10 millimeter (mm) in long axis when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam. Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI.
5. Tumor accessible and participant consents to undergo fresh tumor biopsies.
6. Female participants 18 years or older.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
8. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 90 days (or longer, as mandated by local labeling [example, United States Prescribing Information (USPI), Summary of Product Characteristics (SmPC), etc.]) after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
9. Clinical laboratory values as specified below within 4 weeks before the first dose of study drug:

   * Bone marrow reserve consistent with absolute neutrophil count (ANC) >= 1500 per micro liter (/mcL); platelet count >= 100,000/mcL; hemoglobin A1c (HbA1c) less than (<) 6.5 percent (%).
   * Total bilirubin must be less than or equal to (<=) 1.5 * the upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be <= 2.5 * the upper limit of the normal range. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of metastatic disease in liver.
   * Creatinine clearance >= 50 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) based either on Cockcroft-Gault estimate or based on a 12- or 24-hour urine collection.
   * Fasting serum glucose < 130 milligram per deciliter (mg/dL) and fasting triglycerides <= 300 mg/dL.
10. Ability to swallow oral medications, willingness to perform mucositis prophylaxis, and suitable venous access for the study-required blood sampling.
11. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug. Women who are lactating and breastfeeding are not eligible.
2. Previous treatment with any weekly taxane regimen.
3. History of severe hypersensitivity reactions to paclitaxel or any of its excipients.
4. Previous treatment with phosphoinositide 3-kinase (PI3K), serine/threonine-specific protein kinase (AKT), dual PI3K/ mammalian (or mechanistic) target of rapamycin (mTOR) inhibitors, target of rapamycin complex 1/2 (TORC1/2) inhibitors or TORC1 inhibitors.
5. Initiation of treatment with hematopoietic growth factors, transfusions of blood and blood products, or systemic corticosteroids (either intravenous [IV] or oral steroids, excluding inhalers) within 1 week before administration of the first dose of study drug (participants already receiving erythropoietin on a chronic basis for >=4 weeks are eligible).
6. Participants who are taking proton pump inhibitors (PPIs) within 7 days of the first dose of study drug or who require treatment with PPIs throughout the trial or those who are taking H2 receptor antagonists within 24 hours of the first dose of study drug.
7. A prothrombin time (PT) or activated partial thromboplastin time (aPTT) above the ULN or a history of a coagulopathy or bleeding disorder.
8. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
9. Sensory or motor neuropathy >= Grade 2.
10. Central nervous system (CNS) metastasis, endometrial leiomyosarcoma, or endometrial stromal sarcoma.
11. Manifestations of malabsorption due to prior gastrointestinal surgery, gastrointestinal disease, or for some other reason that may alter the absorption of sapanisertib or MLN1117. In addition, participants with enteric stomata are also excluded.
12. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active CNS disease, active infection, or any other condition that could compromise participation of the participant in the study.
13. Known human immunodeficiency virus infection.
14. History of any of the following within the last 6 months before administration of the first dose of study drug:

    * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures.
    * Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures.
    * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation, or ventricular tachycardia).
    * Placement of a pacemaker for control of rhythm.
    * New York Heart Association Class III or IV heart failure.
    * Pulmonary embolism.
15. Significant active cardiovascular or pulmonary disease before administration of the first dose of study drug, including:

    * Uncontrolled hypertension (that is, either systolic blood pressure > 180 millimeter of mercury [mm Hg] or diastolic blood pressure > 95 mm Hg).
    * Pulmonary hypertension.
    * Uncontrolled asthma or oxygen saturation < 90% by arterial blood gas analysis or pulse oximetry on room air.
    * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention; or history of valve replacement.
    * Medically significant (symptomatic) bradycardia.
    * History of arrhythmia requiring an implantable cardiac defibrillator.
    * Baseline prolongation of the rate-corrected QT interval (QTc; example, repeated demonstration of QTc interval > 480 millisecond [ms], or history of congenital long QT syndrome, or torsades de pointes).
16. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
17. Participants with endometrioid histology and histologically confirmed expression of estrogen receptors (ER) and/or progesterone receptors (PgR) who have not received prior endocrine therapy and for whom endocrine therapy is currently indicated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 241 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (78):
- United States (21):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arizona Cancer Center, Phoenix, Arizona
  - Marin Cancer Care, Greenbrae, California
  - University of California San Diego Medical Center, La Jolla, California
  - University of California at San Francisco (PARENT), San Francisco, California
  - Stanford School of Medicine, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Augusta University, Augusta, Georgia
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Westwood, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - NYU Langone Medical Center Clinic, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (7):
  - St George Hospital, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Sunshine Hospital, Footscray, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria
- Belgium (5):
  - UZ Antwerpen, Edegem, Antwerpen
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Site Sart Tilman, Liège
  - GasthuisZusters Antwerpen Sint-Augustinus, Wilrijk
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Clinic, Hamilton, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM Hopital Notre-Dame, Montreal, Quebec
- Germany (5):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum, Berlin
- Italy (10):
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Forli - Cesena
  - Spedali Civili di Brescia, Brescia
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Istituto Tumori Napoli Fondazione G. Pascale, Napoli
  - Azienda Unita Sanitaria Locale di Ravenna, Ravenna
  - Istituto Nationale Tumori Regina Elena, Roma
  - Universita degli Studi di Roma "La Sapienza" - Umberto I Policlinico di Roma, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Netherlands (5):
  - Maastricht Universitair Medisch Centrum, Maastricht, Limburg
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Erasmus Medisch Centrum Daniel den Hoed, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Norway (3):
  - Haukeland universitetssykehus, Kvinneklinikken, Bergen
  - Radiumhospitalet, Oslo
  - Stavanger University Hospital, Stavanger
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Instituto Valenciano de Oncologia IVO, Valencia
- United Kingdom (9):
  - Bristol Haematology and Oncology Centre, Bristol, Avon
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - University College London Hospitals, London, Greater London
  - Royal Marsden Hospital, London, Greater London
  - Hammersmith Hospital, London, Greater London
  - The Christie, Manchester, Greater Manchester
  - Royal Marsden Hospital, Sutton, Surrey
  - University Hospital Coventry, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Han SN, Oza A, Colombo N, Oaknin A, Raspagliesi F, Wenham RM, Braicu EI, Jewell A, Makker V, Krell J, Alia EMG, Baurain JF, Su Z, Neuwirth R, Vincent S, Sedarati F, Faller DV, Scambia G. A randomized phase 2 study of sapanisertib in combination with paclitaxel versus paclitaxel alone in women with advanced, recurrent, or persistent endometrial cancer. Gynecol Oncol. 2023 Nov;178:110-118. doi: 10.1016/j.ygyno.2023.09.013. Epub 2023 Oct 14. PMID 37839313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 60 investigative sites in Australia, Belgium, Germany, Italy, Netherlands, Norway, Spain, United Kingdom, Canada and the United States from 01 April 2016 to 30 October 2020.
Pre-assignment Details: The female participants with a diagnosis of endometrial carcinoma were enrolled and randomized into 1:1:1:1 ratio to receive single agent paclitaxel, paclitaxel in combination with sapanisertib, single agent sapanisertib or sapanisertib in combination with MLN1117.
Groups:
- Paclitaxel 80 mg/m^2: Paclitaxel 80 milligrams per square meter (mg/m^2), IV, injection, weekly on Days 1, 8, and 15 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was 13.00 weeks).
- Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg: Paclitaxel 80 mg/m^2, IV, injection, weekly on Days 1, 8, and 15 of a 28-day cycle along with sapanisertib 4 milligrams (mg), capsule, orally on Days 2-4, 9-11, 16-18, and 23-25 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was 20.14 and 18.50 weeks).
- Sapanisertib 30 mg: Sapanisertib 30 mg, capsule, orally, once weekly on Days 1, 8, 15, and 22 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was 6.14 weeks).
- Sapanisertib 4 mg + MLN1117 200 mg: Sapanisertib 4 mg, capsule, orally and MLN1117 200 mg, capsule, orally on Days 1-3, 8-10, 15-17, and 22-24 of a 28-day cycle until disease progression, unacceptable toxicity, or withdraw consent (the median exposure was 7.43 weeks).
Period: Overall Study
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Started | 90 | 90 | 41 | 20
Started | 90 | 90 | 41 | 20
Completed | 18 | 20 | 3 | 2
Completed | 18 | 20 | 3 | 2
Not Completed | 72 | 70 | 38 | 18
Not completed — Death | 58 | 59 | 30 | 16
Not completed — Lost to Follow-up | 4 | 3 | 0 | 1
Not completed — Site Terminated by Sponsor | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 8 | 1
Not completed — Reason not Specified | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg | Total
Number analyzed (Participants) | 90 | 90 | 41 | 20 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.14) | 64.4 (7.63) | 64.0 (6.99) | 62.0 (10.20) | 63.9 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 90 | 41 | 20 | 241
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 4 | 15
  Not Hispanic or Latino | 84 | 80 | 37 | 15 | 216
  Unknown or Not Reported | 3 | 5 | 1 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 77 | 78 | 37 | 18 | 210
  Black or African American | 3 | 4 | 0 | 1 | 8
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Asian | 6 | 3 | 1 | 1 | 11
  Other | 0 | 2 | 2 | 0 | 4
  Not Reported | 3 | 3 | 0 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 5 | 6 | 3 | 2 | 16
  Belgium | 5 | 10 | 2 | 3 | 20
  Germany | 6 | 4 | 1 | 0 | 11
  Italy | 14 | 22 | 9 | 4 | 49
  Netherlands | 2 | 3 | 0 | 0 | 5
  Norway | 3 | 1 | 1 | 0 | 5
  Spain | 10 | 7 | 5 | 6 | 28
  United Kingdom | 9 | 4 | 6 | 2 | 21
  Canada | 15 | 10 | 2 | 0 | 27
  United States | 21 | 23 | 12 | 3 | 59
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is number of participants with data available for height at Baseline.
  cm
    number analyzed (Participants) | 87 | 82 | 41 | 20 | 230
    (all) | 160.60 (6.335) | 160.23 (5.798) | 159.01 (6.471) | 162.67 (5.854) | 160.36 (6.16)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is number of participants with data available for weight at Baseline.
  kg
    number analyzed (Participants) | 87 | 84 | 41 | 20 | 232
    (all) | 73.29 (18.783) | 72.13 (18.433) | 75.35 (17.969) | 71.81 (18.613) | 73.11 (18.418)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in months from the date of randomization to the date of first documentation of progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST v1.1, PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to approximately 30 months
Population: ITT population included all randomized participants. For a participant who had not progressed and was last known to be alive, PFS was censored at the last response assessment that is stable disease (SD) or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Number analyzed (Participants) | 90 | 90 | 41 | 20
months | 3.7 [2.3 to 4.5] | 5.6 [3.8 to 6.2] | 2.1 [1.9 to 3.5] | 2.0 [1.5 to 3.3]
Statistical Analysis 1: Comparison: Paclitaxel 80 mg/m^2 vs Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg; Test type: Superiority; p = 0.178, Stratified Log-rank Test — The p-value was obtained using stratified log-rank test with histological subtype, lines of prior chemotherapy and prior taxane therapy (original stratification values); Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.58 to 1.12] — The hazard ratio was obtained using a stratified Cox proportional hazard model adjusted for histological subtype, lines of prior chemotherapy and prior taxane therapy. A hazard ratio of <1 was considered statistically significant
Statistical Analysis 2: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 30 mg; Test type: Superiority; p = 0.092, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.85, 95% CI 2-sided [1.19 to 2.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 4 mg + MLN1117 200 mg; Test type: Superiority; p = 0.147, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.57, 95% CI 2-sided [1.47 to 4.49] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (Up to approximately 54 months)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Number analyzed (Participants) | 87 | 86 | 41 | 20
Participants | 87 | 86 | 41 | 20

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time in months from the date of randomization to the date of death.
Time Frame: Up to approximately 54 months
Population: ITT population included all randomized participants. Participants without documentation of death at the time of analysis were censored at the date last known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Number analyzed (Participants) | 90 | 90 | 41 | 20
months | 12.7 [9.8 to 19.6] | 13.8 [9.9 to 19.1] | 12.5 [9.0 to 15.7] | 11.1 [2.7 to 17.5]
Statistical Analysis 1: Comparison: Paclitaxel 80 mg/m^2 vs Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg; Test type: Superiority; p = 0.968, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.72 to 1.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 30 mg; Test type: Superiority; p = 0.145, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.50, 95% CI 2-sided [0.95 to 2.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 4 mg + MLN1117 200 mg; Test type: Superiority; p = 0.243, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.87 to 2.73] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP is defined as the time in months from the date of randomization to the date of first documentation of progression. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 30 months
Population: ITT population included all randomized participants. For a participant who has not progressed, TTP was censored at the last response assessment that is SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Number analyzed (Participants) | 90 | 90 | 41 | 20
months | 3.7 [2.5 to 5.4] | 5.7 [3.8 to 7.2] | 2.3 [1.9 to 4.2] | 2.2 [1.8 to 3.7]
Statistical Analysis 1: Comparison: Paclitaxel 80 mg/m^2 vs Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg; Test type: Superiority; p = 0.170, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.57 to 1.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 30 mg; Test type: Superiority; p = 0.224, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.67, 95% CI 2-sided [1.04 to 2.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 4 mg + MLN1117 200 mg; Test type: Superiority; p = 0.244, Stratified Log-rank Test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.28, 95% CI 2-sided [1.32 to 3.96] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a best response of a complete response (CR) or partial response (PR). Per RECIST v1.1, CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Up to 30 months
Population: Safety population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Number analyzed (Participants) | 87 | 86 | 41 | 20
percentage of participants | 18.4 | 24.4 | 4.9 | 0
Statistical Analysis 1: Comparison: Paclitaxel 80 mg/m^2 vs Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg; Test type: Superiority; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.66 to 2.90] — The odds ratio and 95% confidence intervals were obtained using a stratified Cochran-Mantel-Haenszel (CMH) model with histological subtype, lines of prior chemotherapy and prior taxane therapy (original stratification values)
Statistical Analysis 2: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 30 mg; Test type: Superiority; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.04 to 1.14] — The odds ratio and 95% confidence intervals were obtained using a stratified CMH model with histological subtype, lines of prior chemotherapy and prior taxane therapy (original stratification values)
Statistical Analysis 3: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 4 mg + MLN1117 200 mg; Test type: Superiority; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — [estimate comment as in outcome 5, analysis 2]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with CR or PR or SD (SD of any duration). Per RECIST v1.1, CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 30 months
Population: Safety population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Number analyzed (Participants) | 87 | 86 | 41 | 20
percentage of participants | 57.5 | 80.2 | 34.1 | 35.0
Statistical Analysis 1: Comparison: Paclitaxel 80 mg/m^2 vs Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg; Test type: Superiority; Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.53 to 5.96] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 30 mg; Test type: Superiority; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.18 to 0.86] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 4 mg + MLN1117 200 mg; Test type: Superiority; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.15 to 1.21] — [estimate comment as in outcome 5, analysis 2]

7. Secondary Outcome: Clinical Benefit Rate (CBR) at Week 16 (CBR-16)
Description: CBR-16 is defined as the percentage of participants who achieved CR or PR of any duration or have SD with a duration of at least 16 weeks. Per RECIST v1.1, CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Week 16
Population: Safety population included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
Number analyzed (Participants) | 87 | 86 | 41 | 20
percentage of participants | 36.8 | 51.2 | 17.1 | 5.0
Statistical Analysis 1: Comparison: Paclitaxel 80 mg/m^2 vs Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg; Test type: Superiority; Odds Ratio (OR) = 2.62, 95% CI 2-sided [0.89 to 7.67] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 30 mg; Test type: Superiority; Odds Ratio (OR) = 0.15, 95% CI 2-sided [0.05 to 0.51] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Paclitaxel 80 mg/m^2 vs Sapanisertib 4 mg + MLN1117 200 mg; Test type: Superiority; Odds Ratio (OR) = 0.07, 95% CI 2-sided [0.01 to 0.67] — [estimate comment as in outcome 5, analysis 2]

ADVERSE EVENTS:
Time Frame: Up to the end of study (approximately up to 54 months)
Description: At each visit investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of relation to study treatment. All-cause mortality:ITT population(n= 90,90,41,20). Serious and other(non-serious) AEs:Safety population.
Arm/Group | Paclitaxel 80 mg/m^2 | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg | Sapanisertib 30 mg | Sapanisertib 4 mg + MLN1117 200 mg
All-Cause Mortality (participants affected / at risk) | 58/90 | 59/90 | 30/41 | 16/20
Serious Adverse Events (participants affected / at risk) | 23/87 | 47/86 | 14/41 | 7/20
Other Adverse Events (participants affected / at risk) | 85/87 | 86/86 | 41/41 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel 80 mg/m^2 (N=87) | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg (N=86) | Sapanisertib 30 mg (N=41) | Sapanisertib 4 mg + MLN1117 200 mg (N=20)
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Discoloured vomit (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 3 | 3 | 1 | 1
Fatigue (General disorders) | 0 | 2 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 3 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Waist circumference increased (Investigations) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel 80 mg/m^2 (N=87) | Paclitaxel 80 mg/m^2 + Sapanisertib 4 mg (N=86) | Sapanisertib 30 mg (N=41) | Sapanisertib 4 mg + MLN1117 200 mg (N=20)
Nausea (Gastrointestinal disorders) | 29 | 53 | 30 | 16
Diarrhoea (Gastrointestinal disorders) | 31 | 48 | 15 | 13
Vomiting (Gastrointestinal disorders) | 20 | 24 | 31 | 15
Constipation (Gastrointestinal disorders) | 25 | 20 | 14 | 5
Abdominal pain (Gastrointestinal disorders) | 13 | 22 | 6 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 22 | 10 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 13 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 5 | 13 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 10 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 8 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 5 | 6 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 4 | 3 | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 5 | 2 | 1 | 0
Fatigue (General disorders) | 39 | 40 | 18 | 7
Asthenia (General disorders) | 7 | 26 | 9 | 10
Pyrexia (General disorders) | 12 | 13 | 5 | 4
Oedema peripheral (General disorders) | 18 | 10 | 2 | 1
Peripheral swelling (General disorders) | 5 | 5 | 0 | 2
Chills (General disorders) | 1 | 5 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 16 | 33 | 20 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 17 | 15 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 19 | 7 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 11 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 8 | 6 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 12 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 8 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 6 | 4 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 6 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 32 | 48 | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 10 | 19 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 8 | 12 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 12 | 22 | 3 | 0
Dysgeusia (Nervous system disorders) | 10 | 15 | 6 | 2
Headache (Nervous system disorders) | 4 | 13 | 6 | 1
Dizziness (Nervous system disorders) | 3 | 14 | 3 | 2
Paraesthesia (Nervous system disorders) | 6 | 9 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 8 | 0 | 0
Tremor (Nervous system disorders) | 2 | 5 | 3 | 1
Taste disorder (Nervous system disorders) | 2 | 6 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 25 | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 19 | 8 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 11 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 27 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 17 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 11 | 6 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 8 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 2 | 1 | 0
Weight decreased (Investigations) | 2 | 17 | 7 | 3
Gamma-glutamyltransferase increased (Investigations) | 6 | 9 | 5 | 0
Alanine aminotransferase increased (Investigations) | 5 | 7 | 1 | 6
Aspartate aminotransferase increased (Investigations) | 3 | 7 | 2 | 6
Neutrophil count decreased (Investigations) | 8 | 9 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 6 | 3 | 4
White blood cell count decreased (Investigations) | 5 | 9 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 5 | 4 | 0
Platelet count decreased (Investigations) | 2 | 2 | 1 | 2
Protein total decreased (Investigations) | 1 | 1 | 3 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 22 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 11 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 16 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 10 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 9 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 9 | 19 | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 5 | 2 | 0
Sinusitis (Infections and infestations) | 5 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 17 | 1 | 1
Anxiety (Psychiatric disorders) | 3 | 7 | 3 | 1
Depression (Psychiatric disorders) | 3 | 3 | 5 | 0
Hypertension (Vascular disorders) | 9 | 5 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 5 | 0 | 1
Hypotension (Vascular disorders) | 2 | 6 | 0 | 0
Haematuria (Renal and urinary disorders) | 7 | 8 | 0 | 0
Dysuria (Renal and urinary disorders) | 5 | 6 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 5 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 6 | 3 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 6 | 4 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 4 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT02725268/Prot_001.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT02725268/SAP_000.pdf